CLINICAL TRIAL: NCT03064022
Title: Preterm Infant Multicentre Growth Study
Acronym: PreMGS
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Canadian Foundation for Dietetic Research (CFDR) (Other); Saskatchewan Health Authority - Regina Area (Other); Tufts University (Other)
Responsible Party: Sponsor
Other Study IDs: REB15-2594
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2019-04

CONDITIONS: Preterm Infant
Keywords: weight gain; head circumference; length; neurodevelopment; overweight
MeSH Terms: conditions — Premature Birth; Weight Gain; Overweight | interventions — Growth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Size < the 3rd or 10th percentiles: Infant size smaller than the 3rd or 10th percentiles relative to the Fenton growth chart for weight or head circumference at discharge from neonatal intensive care
  Interventions: Other: Growth
- Rapid early growth: Rapid early growth will be defined as exceeding birthweight in the first week of life
- Growth velocity calculation methods: We will compare a variety of growth velocity calculation methods used in clinical care and research to compare and assess growth velocity calculation methods
- Size for gestational age: Small size for gestational age

INTERVENTIONS:
Other: Growth — Some preterm infants grow at higher rates than others
  Groups: Size < the 3rd or 10th percentiles

SUMMARY:
The purpose of this study is to improve health professionals understanding of preterm infant growth patterns, and to determine if early growth patterns predict risks of adverse metabolic and cognitive outcomes.

DETAILED DESCRIPTION:
The purpose of this study is:

To improve health professionals understanding of preterm infant growth patterns, and to determine if growth patterns (rapid early growth in the first 2 weeks of life, weight less than the 10th percentile at the time of discharge) predict risks of adverse metabolic outcomes (measured as overweight at age 3) once the following variables are controlled for: size at birth (z-score), neonatal morbidities, social determinants of health, and nutritional adequacy in the neonatal intensive care unit (NICU).

To assess diagnostic accuracy of 36-week anthropometric weight, length and head circumference <10th and <3rd percentiles to predict preterm infant cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* < 32 weeks gestational age at birth

Exclusion Criteria:

* infants who had congenital anomalies or those who died prior to discharge

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants
Sampling Method: Non-Probability Sample
Enrollment: 1275 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Neurodevelopment | Twenty-one months of age
  Neurodevelopment (Bayley scale scores II and III), diagnoses of cerebral palsy, or other neurologic impairments) measured

SECONDARY OUTCOMES:
Overweight | Three years of age
  Overweight will be defined as body mass index
Growth patterns | From birth to 50 weeks post-menstrual age
  Growth patterns of preterm infants relative to the Fenton growth chart

CONTACTS AND LOCATIONS:
Overall Officials: Tanis Fenton, PhD RD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Cumming School of Medicine, Calgary, Alberta
  - Regina Qu'Appelle Health Region, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fenton TR, Nasser R, Eliasziw M, Kim JH, Bilan D, Sauve R. Validating the weight gain of preterm infants between the reference growth curve of the fetus and the term infant. BMC Pediatr. 2013 Jun 11;13:92. doi: 10.1186/1471-2431-13-92. PMID 23758808
- [Result] Fenton TR, Senterre T, Griffin IJ. Time interval for preterm infant weight gain velocity calculation precision. Arch Dis Child Fetal Neonatal Ed. 2019 Mar;104(2):F218-F219. doi: 10.1136/archdischild-2018-314843. Epub 2018 Jul 11. PMID 29997166
- [Result] Fenton TR, Griffin IJ, Hoyos A, Groh-Wargo S, Anderson D, Ehrenkranz RA, Senterre T. Accuracy of preterm infant weight gain velocity calculations vary depending on method used and infant age at time of measurement. Pediatr Res. 2019 Apr;85(5):650-654. doi: 10.1038/s41390-019-0313-z. Epub 2019 Jan 25. PMID 30705399
- [Derived] Fenton TR, Nasser R, Creighton D, Elmrayed S, Tang S, Gillis C, Alshaikh B. Critical examination of relationships between early growth and childhood overweight in extremely preterm infants. J Perinatol. 2021 Dec;41(12):2774-2781. doi: 10.1038/s41372-021-01182-8. Epub 2021 Aug 17. PMID 34404924
- See also: Fenton preterm growth chart webpage — http://ucalgary.ca/fenton